CLINICAL TRIAL: NCT01490437
Title: A Prospective Phase 2 Study of PEmetrexed in Combination With Cisplatin in Patients With Advanced UrotheLIal CAnceR
Brief Title: Pemetrexed and Cisplatin in Advanced Urothelial Carcinoma
Acronym: PECULIAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOSG-AMC-0804
Record Dates: First submitted 2011-12-06; First posted 2011-12-13 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Urothelial Carcinoma
Keywords: Advanced urothelial carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Pemetrexed; Cisplatin; Dexamethasone; Absorptiometry, Photon; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PemCis (Experimental): Pemetrexed plus Cisplatin
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Dexamethasone; Drug: Vitamins

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV over 10 minutes on D1 every 3 weeks
  Other Names: Alimta
Drug: Cisplatin — Cisplatin 70 mg/m2 IV over 60 minutes on D1 every 21 days
  Other Names: cisplan
Drug: Dexamethasone — Dexamethasone 4 mg bid PO from D-1 to D2 every 3 weeks
  Other Names: Dexa
Drug: Vitamins — Folic acid 350 ug - 600 ug daily from D-7 daily vitamin B12 1,000 ug every 9 weeks from D-7

SUMMARY:
Pemetrexed has demonstrated a favorable response with minimal toxicity when used as single agent as first-line and second-line treatment for advanced urothelial carcinoma. The response rates were 32% and 28% for the first-line and second-line setting, respectively. Cisplatin is one the most active chemotherapeutic agents in urothelial cancer, frequently used as combination chemotherapy such as GP (gemcitabine plus cisplatin) or MVAC (methotrexate, vinblastine, adriamycin, and cisplatin).

Pemetrexed and cisplatin showed favorable activity profile in advanced non-small cell lung cancer with highly favorable toxicity profile.

This study is to assess the efficacy and safety of pemetrexed plus cisplatin in advanced urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of urothelial (transitional cell) carcinoma with the exception of micropapillary subtype
* Patients must have recurrent disease (locally advanced or metastatic) that is not amenable to local therapy or newly diagnosed distant metastatic disease
* Measurable disease defined by RECIST v.1.0
* ECOG performance status of 2 or better
* Adequate organ and bone marrow function defined as

Exclusion Criteria:

* Other tumor type than urothelial carcinoma
* Presence or history of CNS metastasis
* Prior systemic chemotherapy or immunotherapy (but prior local intravesical chemotherapy or immunotherapy was allowed. And recurrent disease after adjuvant or neoadjuvant cisplatin-based systemic chemotherapy is allowed if the last chemotherapy was administered 1 year or more before the patient enrollment.)
* Presence of second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Peripheral sensory neuropathy grade 2 or worse
* Other serious illness or medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 12 months
  Based on RECIST v.1.0

SECONDARY OUTCOMES:
Progression-free survival | 12 months
Overall survival | 12 months
Safety | 8 months
  Based on NCI CTCAE v.3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi YJ, Lee SH, Lee JL, Ahn JH, Lee KH, You D, Hong B, Hong JH, Ahn H. Phase II study of pemetrexed in combination with cisplatin in patients with advanced urothelial cancer: the PECULIAR study (KCSG 10-17). Br J Cancer. 2015 Jan 20;112(2):260-5. doi: 10.1038/bjc.2014.591. Epub 2014 Nov 27. PMID 25429526